CLINICAL TRIAL: NCT04001569
Title: Phase1b/2 Study of AZD8186 in Combination With Paclitaxel in Patients With Advanced Gastric Cancer
Brief Title: AZD8186 and Paclitaxel in Advanced Gastric Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Keun-Wook Lee, Professor, Seoul National University Bundang Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KCSG-ST18-20
Record Dates: First submitted 2019-06-23; First posted 2019-06-28 (Actual); Last update posted 2019-06-28 (Actual); Status verified 2019-06

CONDITIONS: Solid Tumor; Stomach Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — AZD8186; Paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AZD8186 in combination with paclitaxel (Experimental)
  Interventions: Drug: AZD8186 in combination with paclitaxel

INTERVENTIONS:
Drug: AZD8186 in combination with paclitaxel — Phase 1b is planned for a 4-stage dose level and the traditional 3+3 design is applied. The RP2D will be determined based on the MTD and toxicity profiles.
  In phase 2 part, RP2D from the phase 1b part will be applied.
  * AZD8186 ( )mg po bid, 5 days on, 2 days off
  * Paclitaxel ( )mg/m² on D1,8,15 every 4 weeks

SUMMARY:
AZD8186 is an orally-dosed, selective Phosphatidylinositol 3-kinase (PI3K) β/δ inhibitor that binds to PI3Kβ and PI3Kδ, and inhibits kinase activity and downstream pathways in vitro and in vivo. AZD8186 has shown significant anti-tumor activity in PTEN-deficient preclinical models, including prostate, triple negative breast cancer, squamous lung and germinal center diffuse large B-cell lymphoma models. PTEN deficiency is reported in approximately 20% of patients with gastric cancer and in 35-48% of those with human epidermal growth factor receptor 2(HER2)-positive gastric cancer. To date, there have been no clinical trials with AZD8186 alone or in combination with paclitaxel in advanced gastric cancer. Therefore, it is very important to conduct clinical trials of combination therapy of AZD8186 and paclitaxel in patients with metastatic/recurrent gastric cancer who have failed previous therapy, and to identify the clinical factors and biomarkers that predict effects of the combination therapy.

The purpose of the study is to define the maximal tolerated dose (MTD) and recommended phase 2 dose (RP2D) of paclitaxel and AZD8186 combination therapy in patients with advanced tumors and to evaluate the efficacy of paclitaxel and AZD8186 combination therapy as a second-line therapy in patients with advanced gastric cancer with PTEN aberrations. This study is divided into Phase 1b and Phase 2.

ELIGIBILITY:
Inclusion Criteria:

1. Have the willingness to sign a written informed consent document prior to any study specific procedures
2. Age ≥ 19 years of male and female
3. At each phase of the trial, subjects who meet the following requirements in the appropriate phase will be enrolled.

   A. Phase 1b: Subjects with a histologically confirmed metastatic solid tumor that have progressed after treatment with approved therapies or for which there is no standard effective therapy available.

   B. Phase 2b: Subjects with histologically confirmed locally advanced or metastatic gastric cancer that have progressed after treatment with first-line fluoropyrimidine-based chemotherapy, with PTEN loss by immunohistochemistry (IHC), PTEN gene abnormality (PTEN gene deletion or loss of function mutation) or Phosphatidylinositol-4,5-Bisphosphate 3-Kinase Catalytic Subunit Beta(PIK3CB) gene abnormality (amplification or gain of function mutation) identified by next generation sequencing (NGS). If the subject received adjuvant chemotherapy after curative gastric resection and lymph node dissection, adjuvant chemotherapy is considered to be the first-line palliative chemotherapy if the disease recurred during adjuvant chemotherapy or within 6 months after the completion of adjuvant chemotherapy.
4. Patients must have measurable disease based on RECIST 1.1 (Phase 2 part only). Measurable disease will not be required for enrollment in the phase1b part. Patients with evaluable lesion only (without measurable lesion) can be enrolled in the phase 1b part.
5. Eastern Cooperative Oncology Group(ECOG) performance status 0-1
6. Patients must have adequate organ and marrow function as defined below:

   A. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L, B. Hemoglobin ≥ 9.0 g/dL, C. Platelet ≥ 100 x 109/L, D. Aspartate transaminase(AST) and/or alanine transaminase(ALT) ≤ 3 × upper limit of normal (ULN) [Regardless of the presence of liver metastases, only subjects who have AST/ALT ≤ 3 × ULN can be enrolled in phase 1b part; In phase 2 part, subjects with AST and/or ALT ≤ 5 X ULN can be enrolled if they have liver metastases] E. Total bilirubin: ≤ 1 × ULN; Subjects with a bile duct obstruction will be eligible if they meet the criteria after appropriate bile drainage; Patients with Gilbert syndrome should also be registered after confirming that the total bilirubin level is within the normal range through a follow-up screening test F. Serum creatinine clearance >50 milliliter/min
7. Adequate cardiac function with corrected QT interval(QTc) < 470 msec
8. Patients must be able to swallow and retain oral medications
9. Serum β-human chorionic gonadotropin (HCG) test negative within 14 days before the first administration (women of childbearing potential only).
10. Requirements for contraception must be followed.

Exclusion Criteria:

1. Active central nervous system (CNS) lesions (ie, those with radiologically unstable or symptomatic brain lesions). For those who receive radiation or surgical treatment, the subject can be enrolled if the subject is maintained without evidence of CNS disease progression for more than 4 weeks. However, patients with a leptomeningeal metastases are excluded.
2. Treatment with any of the following:

   * Nitrosourea or mitomycin C within 6 weeks of the first dose of study treatment
   * Any cytotoxic chemotherapy from a previous treatment regimen within 14 days. If the subject received an investigational drug from another clinical trial, the subject can be enrolled after 2 weeks of last administration and more than 5 x half-life of the investigational drug. If monoclonal antibody therapy was given, the subject can be enrolled after four weeks after the last dose.
   * Strong or moderate inducers or inhibitors of CYP3A4 within 2 weeks before the first dose of study treatment
   * Radiotherapy with a wide field of radiation within 4 weeks or radiotherapy with a limited field of radiation for palliation within 2 weeks of the first dose of study treatment.
   * Any previous exposure to a Phosphatidylinositol 3-kinase (PI3K) inhibitor (including selective or pan PI3K inhibitors), Akt, mammilian target of rapamycin (mTOR) inhibitors.
3. History of allogeneic bone marrow transplantation or organ transplantation
4. History of another primary cancer (excluding gastric cancer):

   Exceptions are:
   * Adequately treated non-melanoma skin cancer (basal cell or squamous cell carcinoma), curatively treated in situ cancer of the cervix, completely resected thyroid cancer without distant metastasis in which all treatment has been completed (Appropriate wound healing is required prior to clinical trial enrollment)
   * Other curatively treated solid tumors except for gastric cancer with no evidence of disease recurrence at least 36 months before participating in this trial
5. Clinically significant cardiovascular disease including but not limited to:

   * Acute coronary syndrome within the 6 months prior to the initiation of study drug (including myocardial infarction or unstable angina, Coronary Artery Bypass Graft surgery, percutaneous coronary intervention and stenting)
   * Current heart failure or past history of heart failure
   * Current or past history of clinically significant cardiac arrhythmia (eg, complete left bundle branch block, third degree heart block)
   * Any risk factors that prolong QTc or increase the probability of arrhythmia, including medication (eg: heart failure, hypokalemia, congenital long QT syndrome, history of Torsades de Pointes)
6. Persistent uncontrolled hypertension as defined by: systolic >180 mmHg or diastolic >100 mmHg despite medical treatment
7. Seropositivity of HIV, or known active hepatitis B and/or active hepatitis C infection. Hepatitis B carriers may be enrolled if prophylactic use of an antiviral agent with minimal interaction with CYP3A4 is administered to inhibit hepatitis B virus (HBV) activation (eg. Entecavir, adefovir)
8. Impairment of gastrointestinal function or gastrointestinal disorders (eg. untreated ulcerative disorders; uncontrolled nausea, vomiting, or diarrhea; absorption disorder syndrome; small bowel resection; ileostomy). Patients with ileostomy will not allowed to be enrolled, but patients with colostomy can be enrolled to this study.
9. As judged by the Investigator, all other symptoms and associated disease for which the investigator determined that participation in this study is contraindicated (e.g. Infection/inflammation; severe liver dysfunction; bilateral diffuse interstitial lung disease; uncontrolled renal disease; unstable heart and lung disease; hemorrhagic disease; intestinal obstruction; unable to swallow oral pills; social and psychological problems, etc)
10. Pregnant or lactating women.
11. Medical, psychiatric, cognitive, or other conditions that may interfere with the ability of the subject to understand the study information, provide the informed consent, follow the protocol process, or complete the clinical trial
12. Hypersensitivity to paclitaxel

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2019-05-14 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximal tolerated dose | 4 weeks
Recommended phase 2 dose | 4 weeks
Progression-free survival rate | 4 months

SECONDARY OUTCOMES:
Dose-limiting toxicity | 4 weeks
  Dose-limiting toxicity (DLT) assessment will be performed during the first cycle in phase 1b part, and is based on NCI-CTCAE (version 4.0).
Overall survival | 1-year
Progression-free survival | 1-year
Objective response rate | 1-year
Adverse event | 1-year

CONTACTS AND LOCATIONS:
Overall Officials: Keun-Wook Lee, MD. & Ph.D, Principal Investigator — Seoul National University Bundang Hospital
Locations (3):
- South Korea (3):
  - Hallym University Sacred Heart Hospital, Anyang-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Asan Medical Center, Seoul

REFERENCES:
- [Derived] Suh KJ, Ryu MH, Zang DY, Bae WK, Lee HS, Oh HJ, Kang M, Kim JW, Kim BJ, Mortimer PGS, Kim HJ, Lee KW. AZD8186 in Combination With Paclitaxel in Patients With Advanced Gastric Cancer: Results From a Phase Ib/II Study (KCSG ST18-20). Oncologist. 2023 Sep 7;28(9):e823-e834. doi: 10.1093/oncolo/oyad059. PMID 37036671